CLINICAL TRIAL: NCT05405426
Title: TITRE: Trial of Indication-Based Transfusion of Red Blood Cells in ECMO
Brief Title: Trial of Indication-Based Transfusion of Red Blood Cells in ECMO
Acronym: TITRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ravi Thiagarajan, Professor/Division of Cardiovascular Critical Care, Dept. of Cardiology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: W81XWH-22-1-0301
Record Dates: First submitted 2022-05-02; First posted 2022-06-06 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-03

CONDITIONS: Extracorporeal Membrane Oxygenation; Red Blood Cell Transfusion; Organ Failure, Multiple
Keywords: pediatric; children; ECMO; transfusion; neurodevelopment; TITRE
MeSH Terms: conditions — Multiple Organ Failure | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Intervention Model Description: Two independent study arms will be used: indication-based red blood cell transfusion strategy vs. a center-specific standard of care hemoglobin/hematocrit threshold-based red blood cell transfusion strategy
Who Masked: Outcomes Assessor
Masking Description: Adjudicators for the primary endpoint (organ failure assessment score) will be blinded to treatment assignment. Specialists for neurodevelopmental assessment of participants will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indication-based red blood cell transfusion strategy (Active Comparator): Red blood cell transfusion will occur if the center-specific hemoglobin/hematocrit threshold for transfusion is met AND at least one of the following conditions is present: a) moderate or severe bleeding; b) reduced tissue oxygen delivery, defined as serum lactate >5 mmol/L or 2 serum lactate levels > 3 mmol/L measured 2 hours apart; or c) hemoglobin < 8 g/dL or hematocrit < 25%, except for neonates (age =< 28 d) and children with single ventricle congenital heart disease (age < 1 y) RBC transfusion for hemoglobin < 10g/dL or hematocrit <30% is allowed.
  Interventions: Other: Red blood cell transfusion
- Center-specific hemoglobin/hematocrit threshold-based red blood cell transfusion strategy (Other): Red blood cell transfusion will occur according to each study center's standard of care strategy, typically based on a particular hemoglobin threshold or hematocrit threshold. When hemoglobin or hematocrit decrease to the threshold, red blood cell transfusion is administered.
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — The intervention is a strategy for when red blood cell transfusion will be administered (see description of Arms). However, volume of RBC transfused in the two arms is not specified by this study. Red blood cell transfusion strategy for ECMO weaning and decannulation is not specified by this study. Red blood cell transfusion after ECMO decannulation is not specified by this study.

SUMMARY:
TITRE - Trial of Indication-based Transfusion of Red Blood Cells in ECMO, is a multicenter, prospective, randomized clinical trial. The overarching goal of TITRE is to determine whether restricting red blood cell (RBC) transfusion according to an indication-based strategy for those with bleeding and/or deficit of tissue oxygen delivery, compared with transfusion based on center-specific hemoglobin or hematocrit thresholds, can reduce organ dysfunction and improve later neurodevelopment in critically ill children receiving Extracorporeal Membrane Oxygenation (ECMO) support.

DETAILED DESCRIPTION:
Observational studies of children on ECMO have shown an association between large-volume RBC transfusion and mortality. However, the hematocrit (or hemoglobin) level at which optimal tissue oxygen delivery occurs is unknown. TITRE - Trial of Indication-based Transfusion of Red Blood Cells in ECMO, is a prospective, randomized clinical trial to be conducted at 18-20 study sites. The overarching goal of TITRE is to determine whether restricting RBC transfusion according to an indication-based strategy for those with bleeding and/or deficit of tissue oxygen delivery, compared with transfusion based on center-specific hemoglobin or hematocrit thresholds, can reduce organ dysfunction and improve later neurodevelopment in critically ill children receiving ECMO support.

Aim 1: To test whether children < 6 years of age on ECMO support who are randomized to a strategy of indication-based versus center-specific threshold-based RBC transfusion will have greater improvement in organ function.

Aim 2: To test whether survivors among children age < 6 years on ECMO support who are randomized to indication-based compared to center-specific threshold-based RBC transfusion will have better neurodevelopmental outcomes and health-related QOL at one year post-randomization.

Key design features include: Randomization stratified by patient age (neonate:

=< 28d vs. non-neonate) and by diagnosis (CHD vs. other diagnosis); and a target sample size of 228 patients. Endpoints will be evaluated during ECMO, at hospital discharge, and at 3, 6, 9, and 12 months. To ensure trial integrity, the primary outcome (pSOFA: Pediatric Sequential Organ Failure Assessment score) will be adjudicated by an independent committee and neurodevelopmental assessments will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 6 year at ECMO cannulation
2. Veno-arterial (VA) mode of ECMO
3. First ECMO run during the index hospitalization

Exclusion Criteria:

1. Gestationally-corrected age < 37 weeks at the time of ECMO cannulation
2. Veno-venous (VV) mode of ECMO
3. Patients initially started on VV-ECMO and then transitioned to VA ECMO > 18 hours after ECMO cannulation
4. ECMO used for procedural support (ECMO deployed and decannulated in procedural area with no ICU ECMO care) or ECMO duration expected to be < 24 h
5. Limitation of care in place or being discussed
6. Congenital bleeding disorders
7. Hemoglobinopathies
8. Primary Residence outside country of enrollment
9. Concurrent participation in a separate interventional trial that has potential to impact neurodevelopment status of patient. (note that observational non-interventional studies do not qualify the patient for exclusion). This includes a patient already enrolled in TITRE
10. Lack of access to medical records required for calculation of pre-ECMO pSOFA score due to cannulation for ECMO at a non-trial center.
11. Randomization not possible within 36 h following ECMO cannulation (e.g., due to staffing or delays related to communication with participant family)
12. Planned transition to ventricular assist device (VAD) within 48 hours of commencing ECMO.
13. Clinically documented indication for a Red Blood Cell transfusion threshold that differs from the center-specific transfusion threshold (e.g., oncological treatment that limits donor exposure).

Ages: 0 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Baseline-adjusted change in pSOFA (pediatric Sequential Organ Failure Assessment) score | At randomization and at 30 days post-randomization (or up to time of ECMO decannulation if earlier; varies according to patient)
  The pSOFA score ranges from 0 (no organ dysfunction) through 24 (severe dysfunction in all 6 organs assessed). If death occurs during ECMO within 30 days, a score of 24 is assigned.
Bayley Infant Scales of Development, 4th edition (Bayley-4) | One year post-randomization (+/- 2 mo)
  Scales for Cognitive, Language (Expressive and Receptive), Motor (Gross and Fine), and Social-Emotional. For ages 16 days to 42 months. Composite score range is 40 to 160.
  Higher scores indicate better performance.
Wechsler Preschool and Primary Scale of Intelligence (WPPSI - IV) | One year post-randomization (+/-2 mo)
  Index scores include Verbal Comprehension, Visual Spatial, Working Memory, and Full Scale Intelligence Quotient (IQ). Score range is 40 to 160. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Mixed venous oxygen saturation | Daily AM (6 AM - 12 AM), during ECMO (up to 30 days post-randomization, whichever is earlier)
  Oxygen content of blood that returns to the heart after meeting tissue needs
Total volume of blood products administered | 30 days post-randomization (or up to time of ECMO decannulation if earlier; varies according to patient)
  Packed RBC and whole blood, cryoprecipitate, plasma, platelets
Presence vs. absence of hospital-acquired Infection | 30 days post-randomization (up to time of ECMO decannulation if earlier; varies according to patient)
  Nosocomially-acquired infection that is not present or incubating at the time of admission to hospital
Daily renal function | Daily up to 30 days post-randomization (or up to time of ECMO decannulation if earlier; varies according to patient)
  Serum creatinine, blood urea nitrogen (BUN)
Acute kidney injury > stage 2 | 30 days post-randomization (up to time of ECMO decannulation if earlier; varies according to patient)
  Kidney Disease Improving Global Outcomes (KDIGO) definition
Number of ECMO circuit component replacements | At 30 days post-randomization
  Replacement of oxygenator and/or pump
Presence vs. absence of hemolysis | Daily up to 30 days post-randomization (or up to time of ECMO decannulation if earlier; varies according to patient)
  According to plasma hemoglobin values
All-cause mortality | 30 days, in-hospital, and 1 year post-randomization
  Death from any cause
Discharge location | At time of hospital discharge (assessed up to 1 year)
  Home vs. rehabilitation facility
Adaptive Behavior Assessment System-3 (ABAS-3) | 1 year post-randomization (+/- 2 mo)
  Composite scores for overall adaptive functioning (General Adaptive Composite, GAC), Conceptual, Social and Practical domains as well as nine subscales. Higher score indicates better behavior.
Child Behavior Checklist (CBCL) | 1 year post-randomization (+/- 2 mo)
  Parent-report; child minimum age 1.5 years. Higher score indicates worse behavior.
Pediatric Quality of Life Inventory 4.0 (PedsQL 4.0) | 9 months post-randomization (+/- 1 mo)
  Parent-report; child minimum age 2.0 years. Higher score indicates better quality of life.
Pediatric Quality of Life Inventory Cardiac Module | 9 months post-randomization (+/- 1 mo)
  Parent-report; child minimum age 2.0 years. To be completed for participants with a congenital heart disease diagnosis. Higher score indicates better quality of life.
Number of Donor Exposures | Daily up to 30 days post-randomization (or up to time of ECMO decannulation if earlier; varies according to patient)
  Number of Donor Exposures for RBC transfusion
Recannulation for ECMO < 48 hours and < 72 hours after decannulation | From ECMO decannulation hour to 72 hours following ECMO decannulation
  No: of patients recannulated for ECMO within 48 hours and 72 hours post-decannulation
ECMO duration | During Hospitalization: From ECMO cannulation to ECMO decannulation, death, transition to Ventricular Assist Device (VAD) or 365 days post-randomization, whichever is earliest
  ECMO duration in hours: Time period from ECMO cannulation to first successful ECMO decannulation in hours. Time accrued during ECMO for additional ECMO runs (i.e. those cannulated within 36 hours following first decannulation) will be included as total ECMO duration
Duration of mechanical ventilation post-randomization | During Hospitalization: From Randomization to Extubation from Mechanical Ventilation, death, hospital discharge, or 365 days post-randomization, whichever is earliest
  Duration of mechanical ventilation post-randomization in hours: Randomization to first successful extubation from mechanical ventilation hours; for patients with tracheostomy that require mechanical ventilatory support at the time of ICU discharge: time of ICU discharge to compute mechanical ventilation duration.
Occurrence of Seizures | Randomization to Hospital Discharge or 90 days post-randomization, whichever is earliest
  Occurrence of electroencephalographic evidence of seizure prior to hospital discharge or within 90 d post randomization, whichever is earliest
Stroke or Intracranial Hemorrhage during ECMO | Time of ECMO cannulation to ECMO decannulation, death or 30 days post-randomization, whichever occurs first
  Occurrence of brain infarction, intracranial hemorrhage, or ischemic injury during ECMO (composite) confirmed using head ultrasound and Computed Tomography (CT) during ECMO
Stroke or Intracranial Hemorrhage prior to Hospital Discharge | ECMO cannulation to 90 days post-randomization or hospital discharge, whichever occurs first
  Proportion of patients with brain infarction, intracranial hemorrhage, or ischemic injury (composite) confirmed using head ultrasound, CT, or Magnetic Resonance Imaging (MRI) prior to hospital discharge or within 90 d post randomization, whichever is earliest
Pediatric Overall Performance Category (POPC) | Randomization to study completion (completion of 12 month neurodevelopment assessment)
  Pediatric Overall Performance (POPC; score range 0 to 6; Unit: categories on a scale; value: lower is better) at Hospital Discharge, 3, 6, 9, 12 months post-randomization.
Functional Status Score (FSS) | Randomization to study completion (completion of 12 month neurodevelopment assessment)
  Functional Status Score (FSS; score range 6 to 30; Unit: numerical value on a scale; lower is better) at hospital discharge, 3, 6, 9, 12 months post-randomization
ICU Length of Stay among survivors during index hospitalization | ICU Admission to ICU discharge, death or 365 post-randomization, whichever occurs first
  Duration of hospitalization in the ICU among survivors in days during index hospitalization. For ICU readmissions only the only days in the first 2 ICU readmissions will be included
Hospital length of stay among survivors during index hospitalization | Hospital Admission to discharge death, or 365 days post-randomization, whichever occurs first
  Duration of hospitalization among survivors in days during index hospitalization
Pediatric Cerebral Performance Category (PCPC) | Randomization to study completion (completion of 12 month neurodevelopment assessment)
  Pediatric Cerebral Performance Category (POPC; score range 0 to 6; Unit: categories on a scale, lower is better) at Hospital Discharge, 3, 6, 9, 12 months post-randomization.
Number of ICU admissions prior to discharge from index hospitalization among survivors | Index ICU discharge to Hospital discharge or 365 days post-randomization, whichever occurs first
  Number of ICU admissions during index hospitalization. ICU admissions are defined as number of ICU admissions following discharge from the first ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn A. Sleeper, ScD, Principal Investigator — Boston Children's Hospital
Locations (22):
- United States (20):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MUSC Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Health Dallas University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Inova Children's Hospital, Falls Church, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No